CLINICAL TRIAL: NCT07404930
Title: Supplementation With L. Reuteri SGL 01 in Nursing Mothers: Evaluation of the Microbiota in Breast Milk and Intestinal Colonization in Newborns
Brief Title: L. Reuteri SGL 01 in Nursing Mothers: Effects on Milk Microbiota and Neonatal Gut Colonization
Acronym: Reuteri17
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Head of Neonatology unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Reuteri17
Record Dates: First submitted 2026-01-21; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Microbiota; Supplementation; Breastfeeding
Keywords: microbiota; breastfeeding; neonates
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemented group (Active Comparator): Daily oral supplementation with 1 × 10⁹ colony-forming units (CFU) of L. reuteri SGL 01 to breastfeeding mothers
  Interventions: Dietary Supplement: probiotic Lactobacillus reuteri SGL 01
- Non-supplemented group (No Intervention): Breastfeeding mothers who received no supplementation

INTERVENTIONS:
Dietary Supplement: probiotic Lactobacillus reuteri SGL 01 — 5 drops of supplement based on lactic acid bacteria consisting exclusively of Lactobacillus Reuteri SGL 01
  Arms: Supplemented group

SUMMARY:
The Reuteri17 study is a spontaneous, prospective, randomized intervention study designed to evaluate the effects of maternal supplementation with the probiotic Lactobacillus reuteri SGL 01 on the composition of the breast milk microbiota and subsequent intestinal colonization of the newborn.

The protocol involves the enrollment of 20 primiparous mothers of full-term, exclusively breastfed infants. Participants are divided into two groups: the first receives a daily supplement of 5 drops of Reuplus® (equivalent to 1 billion live cultures), while the second serves as a non-supplemented control group.

The effectiveness of the intervention is monitored through two sampling moments: at baseline (T0) and after 30 days of treatment (T1). Specifically, 20 ml samples of breast milk and fecal samples from the newborns are collected. Bacterial DNA is extracted from these biological matrices and analyzed using real-time PCR at the University of Bologna, with the aim of quantifying changes in the microbiota and the transfer of the probiotic strain.

To complete the investigation, mothers are given a nutritional questionnaire to correlate the results with dietary habits. The study aims to confirm that maternal oral supplementation can be an effective strategy for modulating the bacterial heritage of newborns during the first months of life.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women, mothers of full-term infants who are breastfed.
* Written informed consent;
* Age over 18 years.

Exclusion Criteria:

* Drug therapies that are contraindicated for breastfeeding
* Maternal conditions that are contraindicated for breastfeeding
* Neonatal formula milk feeding
* Antibiotic treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in the concentration of Lactobacillus, Bifidobacterium, Clostridium and Bacteroides spp. in maternal milk samples between T0 and T1 | 30 days
  Bacterial DNA was extracted from 2 mL of milk samples, stored at -80 °C after collection, using the QIAamp DNA Mini Kit (Qiagen, West Sussex, UK). Bacterial counts (log CFU/ml milk) were based on rRNA gene copy numbers retrieved from the rRNA copy number database. Mann-Whitney U test was used to compare the concentration of Lactobacillus, Bifidobacterium, Clostridium and Bacteroides spp. in milk samples at T0 and T1 between the study groups. Wilcoxon signed rank test was used to compare the concentration of Lactobacillus, Bifidobacterium, Clostridium and Bacteroides spp. in milk samples between T0 and T1 within each study group. Significance level was set at P <0.05.
Changes in the concentration of Lactobacillus, Bifidobacterium, Clostridium and Bacteroides spp. in neonatal fecal samples between T0 and T1 | 30 days
  Bacterial DNA was extracted from 250 mg of neonatal fecal samples, stored at -80 °C after collection, using the QIAamp DNA Mini Kit (Qiagen, West Sussex, UK). Bacterial counts (log CFU/g feces) were based on rRNA gene copy numbers retrieved from the rRNA copy number database. Mann-Whitney U test was used to compare the concentration of Lactobacillus, Bifidobacterium, Clostridium and Bacteroides spp. in neonatal fecal samples at T0 and T1 between the study groups. Wilcoxon signed rank test was used to compare the concentration of Lactobacillus, Bifidobacterium, Clostridium and Bacteroides spp. in fecal samples between T0 and T1 within each study group. Significance level was set at P <0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Aoubo, Bologna, BO, Italy